CLINICAL TRIAL: NCT06535581
Title: Perfusion Index in the Follow-up of Postoperative Pain; Hypertension Patient Sample
Brief Title: Perfusion Index in the Follow-up of Postoperative Pain
Status: Completed | Type: Observational
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Harun Tolga Duran, M.D., Amasya University
Other Study IDs: E-76988455-050
Record Dates: First submitted 2024-07-26; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Perfusion; Complications
Keywords: perfusion index; postoperative pain; anaesthesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Medical Errors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: hypertension patients
  Interventions: Procedure: surgery patient
- group 2: non hypertension patients
  Interventions: Procedure: surgery patient

INTERVENTIONS:
Procedure: surgery patient — patients with hypertension (group 2) and without (group 1) hypertension. The predictive ability of postoperative pain as a tool for measuring and assessing pain was examined by analysing the relative change in the Perfuston index.

SUMMARY:
Background: The effect of the perfusion index (PI) as an indicator of postoperative pain was investigated. To this end, the presence of the perfusion index in predicting the need for analgesia and its effect in hypertensive patients were investigated. Researher aimed to investigate the change in perfusion index in the prediction of postoperative pain after laparotomic abdominal surgery. As a secondary aim, the results of the relative change in perfusion index in the presence of hypertensive disease were analysed. Methods: A total of 100 patients with ASA 1-3 with or without hypertension who were scheduled to undergo open abdominal surgery between 1 April 2023 and 30 November 2023 were included in the study. The relative variability of visual analogue scale (VAS) and PI in patients receiving postoperative analgesia was examined. The degree of prediction of postoperative pain by these variables after rescue analgesia was investigated. Hypertensive patients were analysed along with other patient groups.

DETAILED DESCRIPTION:
In this prospective randomized single-blind cohort study, postoperative visual analog scale and perfusion index change were examined. Relative changes in VAS and PI were analyzed.

Researher included a total of 100 adult participants with American Society of Anesthesiologists physical statuses ranging from 1 to 3, who were scheduled to undergo laparotomy abdominal surgery under general anesthesia. Exclusion criteria were as follows: Patients with difficult cooperation and heart failure were excluded from the study 2.3Allocation,Randomization On the day of surgery, patients without hypertension disease (Group 1) and those with hypertension disease (Group 2) were separated and taken into surgery. Routine electrocardiography (ECG), pulse oximetry and blood pressure monitoring and pulse oximetry devices (Masimo Corp, Irvine CA, USA) were used to record mean arterial pressure (MAP), PI and pleth variability index (PVI) values at the start of anaesthesia.

The study was conducted at Amasya Sabuncuoğlu Şerefettin Training and Research Hospital and approved by the ethics committee with the number 2023000037-1. All studies were informed about the study and informed consent was given. All patients were routinely given 500 cc of Ringer's lactate solution intravenously in the preoperative period before anaesthesia and taken to the operating room. Written informed consent was obtained from volunteers and included in the study. . All patients received intravenous (IV) hydration with 500 cc of Ringer's lactate after a 6-hour fast. For premedication, midazolam 1 mg IV and pantoprazole 40 mg IV were administered 10 minutes before the operating room. Routine electrocardiography (ECG), pulse oximetry and blood pressure monitoring and pulse oximetry devices (Masimo Corp, Irvine CA, USA) were used to record mean arterial pressure (MAP), PVI values at the start of anaesthesia.

Propofol 2 mg/kg, fentanyl 2 µg/kg and rocuronium 0.6 mg/kg were administered intravenously to induce anaesthesia. Endotracheal intubation was performed after muscle relaxation under deep anaesthesia. Post-induction anaesthesia was maintained with sevoflurane 2%, 50-50% oxygen-air mixture. After surgery, the effect of muscle relaxation was terminated with sugammadex 200 mg and patients were transferred to the post-anaesthesia care unit when sufficient muscle strength was observed. Paracetamol 500 mg iv and tramadol 100 mg iv were administered postoperatively. Postoperative pain was assessed using a VAS. Pain was scored on a 0-10 scale, and a VAS > 6 was considered the pain cut-off point for rescue analgesia. When the patient first arrived at the post-anaesthesia care unit, a VAS 0 value was accepted and scoring was performed every 30 minutes (VAS 30, VAS 60, VAS 90). The corresponding PI 0, PI 90, PVI 0, PVI 90 values were recorded. If VAS>6, morphine 0.05 mg/kg was repeated every 15 minutes until VAS <6 as rescue analgesia. Patients with a modified Aldrete score >8 were observed and referred to the clinical unit. Relative changes in VAS score were calculated during statistical analysis. VAS 1 was taken as the last value measured after rescue analgesia in the post-anaesthesia care unit. The relative change was calculated as ( ΔVAS)=(VAS 0-VAS 1)/(VAS 0). Similarly, relative changes in PI were calculated using the formula ( ΔPI)=(PI 0-PI 1)/(PI 0). These changes were analysed in patients with hypertension (group 2) and without (group 1) hypertension. The predictive ability of postoperative pain as a tool for measuring and assessing pain was examined by analysing the relative change in the Perfuston index.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical statuses ranging from 1 to 3, who were scheduled to undergo laparotomy abdominal surgery under general anesthesia.

Exclusion Criteria:

* Patients with difficult cooperation and heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: laparotomy abdominal surgery under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
PI value | minutes 90
  The correlation between the relative change in PI value and the relative change in VAS value after anesthesia induction and postoperative pain management was investigated.
hypertension patient | minutes 90
  The relative change in PI value and the relative change in VAS value were compared in hypertensive patients and non-hypertensive patients.

SECONDARY OUTCOMES:
complication | minutes 90
  Complications developing in all patients

CONTACTS AND LOCATIONS:
Overall Officials: harun duran, md, Principal Investigator — Amasya University
Locations (1):
- Amasya University Training and Research Hospital, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data sources may be shared depending on the type or plan of the study.

REFERENCES:
- [Background] Bihani P, Pandey A, Jha M, Paliwal N, Jaju R, Solanki R. Comparing Perfusion Index and Visual Analogue Scores for Postoperative Pain Assessment Following Upper Limb Surgeries Under Supraclavicular Brachial Plexus Block: An Observational Study. Cureus. 2024 Mar 4;16(3):e55529. doi: 10.7759/cureus.55529. eCollection 2024 Mar. PMID 38576659
- [Background] Kamel AAF, Medhat MM, Salem DAE, Naby SMA. Effect of perioperative magnesium sulfate and labetalol infusion on peripheral perfusion and postoperative pain in nasal surgery: a randomized controlled trial. Patient Saf Surg. 2022 Aug 19;16(1):27. doi: 10.1186/s13037-022-00336-7. PMID 35986325
- [Background] Elshal MM, Hasanin AM, Mostafa M, Gamal RM. Plethysmographic Peripheral Perfusion Index: Could It Be a New Vital Sign? Front Med (Lausanne). 2021 Oct 1;8:651909. doi: 10.3389/fmed.2021.651909. eCollection 2021. PMID 34660615